CLINICAL TRIAL: NCT00932009
Title: Prevalence and Type Distribution of Genital Human Papillomavirus (HPV) in Tanzanian Men
Brief Title: Prevalence and Type Distribution of Human Papillomavirus (HPV) in Tanzanian Men
Status: Completed | Type: Observational
Sponsor: Danish Cancer Society (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Susanne Kruger Kjaer, Professor, Danish Cancer Society
Other Study IDs: HPV IISP #36113
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Human Papillomavirus Infection
Keywords: Human papillomavirus infection; Tanzanian men; Prevalence
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — cell scrapes from penis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Human papillomavirus: Tanzanian men with HPV and Tanzanian men without

SUMMARY:
The purpose of this study is to determine the prevalence and type distribution of genital human papillomavirus (HPV) infection in Tanzanian men.

DETAILED DESCRIPTION:
STUDY POPULATION The study will be performed in an urban and a rural setting in Tanzania. In the urban setting we aim to include men from different employment categories at larger industries, which potentially have already been identified (Twinga cement, ALAF-Aluminum Company, Bakhresa Food Industry, Simba plastics Industry, and Mohamed Enterprise Food Industry), and in addition we will include men from the College/University environment in Dar es Salaam (Vocational Education Training Dar-es-salaam branch, and Dar-es-salaam Institute of Transport). From the 2002 Census it has been estimated that the population of Dar es Salaam was 2,497,940

The recruitment of men for the study in the rural setting will take place in villages in the Kihaba district and the Bagamoyo district.

Kibaha is one of the 6 districts of the Pwani Region located in Eastern Tanzania. It is the capital of Pwani region. The district is bordered to the North by the Bagamoyo District, to the East by Dar-es-Salaam, to the South by the Kisarawe District and to the West by the Morogoro Region. One of the villages potentially selected for this study is Mlandizi village located in Kibaha district. According to the 2002 Tanzania National Census, the population of the Kibaha District was 132,045 Bagamoyo is also one of the 6 districts of the Pwani Region of Tanzania. It is bordered to the North by the Tanga Region, to the West by the Morogoro Region, to the East by the Indian Ocean and to the South by the Kibaha District. The district capitol is at Bagamoyo. According to the 2002 Tanzania National Census, the population of e.g. the Bagamoyo District was 230,164.

The overall study population in the present investigation will include 2000 men aged 18-60 years. Based on our experience from the recent male study conducted in Denmark and also on the experience obtained in the female study in Tanzania, we will establish a study team that will travel to the different study sites and obtain the penile samples, do interviews, and be responsible for the HIV counseling at the respective study site. The study team will consist of a male doctor to take the penile swabs, two male study assistants to do the interviews, and one HIV counselor. We will also employ a Danish researcher who will work together with the Tanzanian doctor and the rest of the study team in the data collection and entry of the data. Dr. Crispen Kahesa, who was also involved in our study of HPV infection in Tanzanian women, and the Danish researcher will collaborate in the day-to-day conduct of the study with the supervision/assistance of Dr Julius Mwaiselage on a weekly basis and with Professor Susanne Krüger Kjær. Before initiation of the study, the Danish part of the team from the Danish Cancer Society will teach the investigating team to take the penile swabs so that it will be done the same way as it was done in the recent Danish male study.

DATA COLLECTION We have chosen an HPV strategy which matches the strategy we are using in the female Tanzanian study and previously have used in our Danish male study, namely initial testing with HC2 followed by genotyping of the samples positive for HC2 high-risk (HR) types and/ or low-risk (LR) types.

HPV DNA prevalence: HPV samples will be obtained by rubbing a moist cotton swab on glans penis (including sulcus coronarius and underneath preputium), the penile shaft, scrotum and perineum following a loosening of the cells with a nail file. This procedure is adapted from the Merck male clinical studies. We have previously documented that this technique is useful for obtaining HPV samples among men (Morré et al., 2000; Morré et al., 2002; Kjær et al. 2005), and most recently, we have included more than 2,500 men from Danish military barracks in a study assessing the presence of HPV DNA and HPV type distribution in Danish men. The HPV samples from the Tanzanian men will be sent with currier to Prof. Iftners laboratory in Germany where they will be tested for HPV by means of the Hybrid Capture 2 (HC2) method (Digene), low-risk and high-risk probes.

HPV type distribution: HPV genotyping will be performed using Papillocheck - a DNA-Chip analysis for the type-specific identification of 18 high-risk and 6 low-risk types of HPV. Alternatively if funding allows it, we will use a reverse hybridization line probe assay test (LiPa test) from Innogenetics (which is more expensive, but is slightly more sensitive than the Papillocheck test, and another advantage is that we have used this test in our Danish HPV study of 2,500 men). The testing strategy will be to genotype all HC2 positive (HR positive and/or LR positive) samples.

Assessment of HIV status: An HIV test will be offered to all men enrolled in the study and performed taking into account the individual person's wish to be tested and informed about their HIV status. HIV antibody presence in whole blood samples will be assessed following the WHO approved HIV serial testing algorithm. Initially, the Bioline HIV-1/2 immunodetection is used, and is subsequently followed by Determine HIV-1/2 test in order to confirm Bioline potentially positive results.

Assessment of risk factors associated with HPV infection: A structured interview focusing on socio-economic characteristics, circumcision status, sexual activity, STI history and knowledge about HPV and the HPV/ cancer relationship, will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* men who are able to understand the information about the study (in writing or oral)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tanzanian men from an urban setting (Dar es Sallam)(factories, University, college)and men from an rural setting (Muhesa, Mwanga, Bagamoyo)
Sampling Method: Non-Probability Sample
Enrollment: 1933 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
HPV infection | At enrollment

SECONDARY OUTCOMES:
HIV infection | At enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Susanne K. Kjaer, Professor MD, Principal Investigator — Inst. of Cancer Epidemiology,Danish Cancer Society
Locations (1):
- Inst. of Cancer Epidemiology, Danish Cancer Society, Copenhagen, Denmark

REFERENCES:
- [Derived] Olesen TB, Munk C, Mwaiselage J, Kahesa C, Rasch V, Frederiksen K, Iftner T, Kjaer SK. Male circumcision and the risk of gonorrhoea, syphilis, HIV and human papillomavirus among men in Tanzania. Int J STD AIDS. 2019 Dec;30(14):1408-1416. doi: 10.1177/0956462419874593. No abstract available. PMID 31795926
- [Derived] Olesen TB, Mwaiselage J, Iftner T, Kahesa C, Rasch V, Frederiksen K, Munk C, Kjaer SK. Risk factors for genital human papillomavirus among men in Tanzania. J Med Virol. 2017 Feb;89(2):345-351. doi: 10.1002/jmv.24627. Epub 2016 Jul 20. PMID 27404999
- [Derived] Olesen TB, Munk C, Christensen J, Andersen KK, Kjaer SK. Human papillomavirus prevalence among men in sub-Saharan Africa: a systematic review and meta-analysis. Sex Transm Infect. 2014 Sep;90(6):455-62. doi: 10.1136/sextrans-2013-051456. Epub 2014 May 7. PMID 24812407
- [Derived] Olesen TB, Iftner T, Mwaiselage J, Kahesa C, Rasch V, Ngoma T, Munk C, Kjaer SK. Prevalence and type distribution of human papillomavirus among 1813 men in Tanzania and the relationship to HIV status. Sex Transm Dis. 2013 Jul;40(7):592-8. doi: 10.1097/OLQ.0b013e31828fcf57. PMID 23965778